CLINICAL TRIAL: NCT02753634
Title: An Innovative Mind-motor Exercise Approach to Osteoarthritis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OA SSE
Record Dates: First submitted 2016-03-22; First posted 2016-04-28 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Square-stepping exercise Intervention (Experimental): Participant attend sessions 2 times per week for 24-weeks at a community location. An instructor demonstrated increasingly difficulty walking or stepping patterns across a gridded mat and participants are asked to try and remember and repeat the patterns. Social engagement is encouraged.
  Interventions: Behavioral: Square-stepping exercise
- Usual care wait-list control group (No Intervention): This group will be invited to participate in square-stepping exercise after final assessments are completed.

INTERVENTIONS:
Behavioral: Square-stepping exercise — Participants are asked to remember and repeat stepping patterns across a gridded mat as shown to them by an instructor.
  Other Names: Mind-motor exercise
  Arms: Square-stepping exercise Intervention

SUMMARY:
Osteoarthritis (OA) is a growing burden in an aging society. There are few proven treatments and hence disability contributes to poor quality of life and direct/indirect costs to society. OA symptoms include both increased pain and reduced mobility. Strength training and aerobic exercise has been shown to improve symptoms in OA; however, the impact of targeted mobility and balance training in patients with osteoarthritis is unclear. The investigators propose a novel, low-impact exercise modality that improves balance and gait. The results of this research project should improve patient options and improve knowledge in OA management.

DETAILED DESCRIPTION:
Patients with OA have increased fall risk, which can lead to reduced mobility and curtailment of daily activities. Patients with OA also show varied and altered mobility in a sit-to-stand test, suggesting that both poor lower limb strength and flexibility need to be addressed with targeted interventions in this population. Altered mobility is also associated with pain in patients with OA. The cause of decreased mobility and increased pain is often a result of body weight. In a 5-year follow-up study, classes of knee OA were identified as being associated with good, moderate or poor outcomes; characteristics of the poor outcomes class included high BMI, worse pain, >2 co-morbidities and avoidance of activities. Avoidance of activities is a particularly important outcome since this could lead to a downward spiral of decreased physical functioning, falls and further avoidance of activities.

Multiple studies have shown that increasing weight from normal to overweight or obese decreases mobility and increases pain in individuals with OA. This is a potential target for non-pharmacological therapies. For example, Messier et al., showed that a diet and exercise intervention designed to promote weight loss in overweight individuals with knee OA, improved knee compressive forces and function, reduced inflammatory marker IL-6, decreased pain and improved physical health-related quality of life over an 18-month period. This study demonstrated the important effects of weight loss and exercise on knee OA for overall health. In a recent review, the evidence was overwhelming regarding the use of exercise as a treatment of knee OA. Specifically, the literature demonstrates that strength training and aerobic exercise can improve outcomes, such as pain reduction and increased function, in patients with OA. Lifestyle interventions should be utilized in OA populations to help reduce pain, improve mobility and reduce fall risk.

Square-Stepping Exercise (SSE) was developed is a low-tech, low-intensity, novel form of exercise developed in Japan. SSE was originally designed to reduce fall risk in older adults. Participants watch, recognize, memorize and follow increasingly more difficult step patterns, which an instructor demonstrates on a 4 by 10 square-patterned mat. In older adult populations, Shigematsu and colleagues have found that SSE improves overall fitness and lower extremity functioning, as well as reduces fall risk, when compared to walking programs or strength and balance training. In combination with Shigematsu's research in Japan in healthy older adults, the investigators are aiming to provide a significant evidence base for SSE internationally and within varied populations, including older adults with osteoarthritis. In collaboration with Dr. Shigematsu, the investigators have executed SSE studies at the Canadian Centre for Activity and Aging in London, ON and most recently in Woodstock, ON. Preliminary evidence from our study at the Canadian Centre for Activity and Aging showed that over a 3-month training period, participants in our Exercise-Intervention (E-I) group (involving mind-motor exercise) improved their total balance scores, compared to an Exercise-Control (E-C) group.

SSE has not been tested in the OA population. This pilot study will add to the literature to determine whether it reduces pain and improves mobility as an additional non-pharmacological treatment for this population.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis

Exclusion Criteria:

* WOMAC less than 4
* Use of braces
* Uncontrolled hypertension
* Significant psychiatric or psychotic disorder
* Not able to attend 75% of sessions
* Any other reason that would prevent participation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
WOMAC Index | Change from baseline to 24-weeks
  self-report of knee pain for osteoarthritis
WOMAC Index | Change from baseline to 12-weeks
  self-report of knee pain for osteoarthritis

SECONDARY OUTCOMES:
30 second Chair stand | change from baseline to 24-weeks
  measures lower limb functional strength
30 second Chair stand | change from baseline to 12-weeks
  measures lower limb functional strength
Timed up and Go test | change from baseline to 24-weeks
  measures functional fitness
Timed up and Go test | change from baseline to 12-weeks
  measures functional fitness
Fullerton Advanced Balance Scale | change from baseline to 24-weeks
  a single scale used to measure static and dynamic balance
Fullerton Advanced Balance Scale | change from baseline to 12-weeks
  a single scale used to measure static and dynamic balance
6 metre walk test | change from baseline to 24-weeks
  measures usual walking speed
6 metre walk test | change from baseline to 12-weeks
  measures usual walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petrella, MD, PhD, Principal Investigator — Western University, Canada

IPD SHARING:
Plan to Share IPD: No